CLINICAL TRIAL: NCT04076007
Title: The Effect of Dietary Nitrate on Blood Pressure, Insulin Resistance and Vascular Function in Type 2 Diabetes
Brief Title: The Effect of Dietary Nitrate on Blood Pressure, Insulin Sensitivity, and Vascular Function in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CRF035
Record Dates: First submitted 2015-06-02; First posted 2019-09-03 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Diabetes; Hypertension
Keywords: nitrate; nitrite; nitric oxide; diabetes; hypertension
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Active Comparator): Nitrate rich beetroot juice (7.5 mmol nitrate in 250mls beetroot juice) once daily.
  Interventions: Dietary Supplement: Beetroot juice
- Placebo (Placebo Comparator): Nitrate depleted beetroot juice (0.002 mmol nitrate in 250 ml beetroot juice) once daily.
  Interventions: Dietary Supplement: Nitrate depleted beetroot juice

INTERVENTIONS:
Dietary Supplement: Beetroot juice
  Arms: Active
Dietary Supplement: Nitrate depleted beetroot juice
  Arms: Placebo

SUMMARY:
Dietary nitrate supplementation has previously been shown to reduce blood pressure in healthy volunteers. The investigators wished to see whether this would be replicated in subjects with type 2 diabetes and age matched healthy controls.

DETAILED DESCRIPTION:
Double blind, randomised placebo control trial, with crossover design comparing the effect of beetroot juice (rich in nitrate) with placebo (nitrate depleted beetroot juice) on blood pressure, endothelial function and insulin sensitivity in subjects with type 2 diabetes. Healthy age matched subjects will have blood pressure measured.

Plan of Investigations: Study outcome measurements.

Blood pressure measured using ambulatory blood pressure monitoring (Spacelabs) for 24 hours.

Urine albumin excretion rate: in overnight samples using standard radioimmunoassay techniques.

Urine nitrate excretion will be used as a measure of adherence, and will be measured using an HPLC assay recently developed at St. Luke's in Professor Winyard's laboratory.

Microvascular endothelial function assessed by iontophoresis of an endothelial -dependent (acetylcholine, ACh) and -independent (sodium nitroprusside, SNP) vasodilator and monitoring of perfusion response using Laser Doppler Perfusion Imaging intra-individual coefficient of variation is 12% for Ach and 18.7% for SNP.

Post-occlusive reactive hyperaemia: A laser Doppler probe will be attached to the inside surface of the forearm or the dorsum of the foot and blood flow will be measured for 5-minutes. Following this, a blood pressure cuff will be rapidly inflated to 200mmHg for 5 minutes to occlude blood flow. At the end of the 4 minute occlusion the cuff will be rapidly deflated and blood flow recorded for 10 minutes post release. This procedure stimulates microvessels to dilate with a consequent increase in blood flow. Analysis involves detailed investigation into the shape of the blood flow curve in order to categorize it into one of 3 options: normal; early dominant peak and early non-dominant peak.

Optical reflectance spectroscopy (ORS) ORS is a non-invasive technique that directly measures both the changes in blood volume and oxygenation of the skin microcirculation. Visible light passing through the skin is attenuated in part by the concentration of oxy- and deoxyhaemoglobin. Assuming the attenuation of light by scattering remains constant, changes in the concentration of oxy- and deoxyhaemoglobin can be calculated from the measured changes in light attenuation at different wavelengths as it travels through the skin.

Skin Maximum Hyperaemia (MH): An area of the dorsal aspect of the right foot and the ventral aspect of the forearm, clear of visible veins or skin lesions, will be heated to a temperature of 42C for 30 minutes with a small brass heater of 1cm in diameter (Moor Instruments, Axminster, Devon, U.K.) and the maximum blood flow response is measured using laser Doppler techniques (single point or laser Doppler perfusion imager. The mean intra-individual coefficient of variation for the measurement of maximum blood flow is 6.6% determined from 2 subjects on 5 separate occasions. Using this technique the investigators have previously observed alterations in skin maximum hyperaemia with type 2 diabetes and in women with a previous history of gestational diabetes.

Near-infrared spectroscopy (NIRS). NIRS is a non-invasive technique that assesses the change in blood volume and oxygenation of the microcirculation in different tissue beds including muscle and brain., it works on the same principles of ORS except that it uses a near-infrared light source rather then visible light. As near-infrared (760 - 840 nm) has a longer wavelength than visible light it scatter less and therefore it has an increased depth of penetration which allows it to assess oxygenation in the muscle or brain where it will be used in relation to our assessment of cognition.

. Insulin sensitivity will be measured at the end of the two treatment phases using a hyper-insulinaemic isoglycaemic clamp (a modified version of the hyperinsulinaemic euglycaemic clamp). A primed, constant rate infusion of soluble insulin (2.0 mukg per min) will be administered for 180min and a variable rate infusion of 20% glucose administered to maintain isoglycaemia . The isoglycaemic set point will be determined by taking the mean of two fasting blood glucose measurements which will be taken on the day of vascular testing and prior to the clamp. The insulin infusion will be prepared in 45 ml of 0.9% NaCI, and 5 ml of the patient's blood to prevent adsorption of insulin to plastic surfaces. At 5 min intervals, 2 ml blood samples will be collected from a dorsal hand vein. During steady state, M is calculated from glucose infusion rate and serum insulin concentration according to a simple mathematical formula.

Flow mediated vasodilatation used as a measure of the production of endothelial nitric oxide to a standard stimulus (shear). As described previously and following consensus guidelines, peripheral vascular endothelium-dependent (i.e. NO-mediated) vasodilatation in response to forearm reactive hyperaemia will be determined by measuring the diameter change of the brachial artery using linear array B-mode ultrasound and automated edge detection software (MIA, Iowa, USA). Reactive hyperaemia will be induced by occlusion of blood flow to the upper forearm using a cuff inflated to 250 mmHg for 5 minutes followed by rapid deflation. Blood flow during reactive hyperaemia will be measured using an Ultrasound Doppler system for the calculation and analysis of the shear-rate stimulus. Vascular endothelium-independent vasodilatation (internal control) will be determined by the brachial artery dilatation to sublingual nitroglycerine (0.4 mg). The intra-individual coefficient of variation for flow mediated dilatation is 8.1%.

VO2 max testing: Static bicycle exercise tests will be performed to determine oxygen uptake kinetics during sub-maximal exercise and maximal oxygen uptake using standard procedures. During the exercise tests, near infra-red spectroscopy will be used to measure the changes in muscle oxy, deoxy and total haemoglobin which accompany exercise.

Cognitive Function Testing: Using the E-prime program (Psychology Software Tools inc) a 30 minute array of cognitive function tests will be devised. The patient will complete these simple tests on a laptop during the acclimatisation period

Plasma Nitrite and Nitrate Deproteinised samples will be analysed for nitrite and nitrate concentration using a Sievers nitric oxide analyser (Sievers NOA 280i, Analytix Ltd, Durham, UK) and a modification of our previous chemiluminescence technique

ELIGIBILITY:
Inclusion Criteria:

* Patients with type II diabetes (as defined by WHO) of at least 5 years duration between the ages of 35-75 known to have blood pressure above 125mmHg systolic and/or 85mmHg diastolic, or who are taking one or two antihypertensive drugs will be invited.

Healthy Control inclusion/exclusion criteria

Inclusion criteria

* Age and sex matched for participants with diabetes
* Not on any regular medication, excluding the oral contraceptive pill
* Able to give informed consent

Exclusion Criteria:

* Patients with significant renal impairment (eGFR<30), uncontrolled hypertension, BMI<25 or >35, are taking regular organic nitrates, nicorandil, glitazones, phosphodiesterase inhibitors, who have had a myocardial infarction or cerebro-vascular event, who smoke, or any other serious medical condition which would interfere with data interpretation or safety will be excluded

Exclusion Criteria

* Antibiotic therapy within the preceding two weeks
* Myocardial infarction or cerebro-vascular event within the preceding three months
* Current smoker
* Any other medical condition which would interfere with data interpretation or safety.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-12; Primary Completion 2012-08 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
24 hour Ambulatory Blood Pressure monitoring after 2 weeks active juice | 2 weeks
  24 hour average systolic, diastolic blood pressure in mm Hg
24 hour Ambulatory Blood Pressure monitoring after 2 weeks placebo juice | 2 weeks
  24 hour average systolic, diastolic blood pressure in mm Hg

SECONDARY OUTCOMES:
Brachial artery Flow mediated vasodilation | After 2 weeks active juice and after 2 weeks placebo juice
  Following release of a downstream occlusive cuff the percentage change from baseline in the diameter of the brachial artery is recorded.
Microvascular response to Iontophoresis of Acetylcholine and Sodium Nitroprusside | After 2 weeks active juice and after 2 weeks placebo juice
  Skin blood flux will be measured following iontophoresis of the vasodilators acetylcholine and sodium nitroprusside. Peak flux and area under the curve measured in arbitrary units of flux.
Peak reactive hyperemia | After 2 weeks active juice and after 2 weeks placebo juice
  Assessment of morphology of peak blood flow following release of occlusion of lower limb arterial supply. Measurements include time to peak blood flow (seconds), time to return to base line flow (seconds) and categorisation of peak shape.
Maximum hyperemia in response to heating | After 2 weeks active juice and after 2 weeks placebo juice
  Peak blood flux in skin in response to localised heating to 42 degrees C
Cognitive function | After 2 weeks active juice and after 2 weeks placebo juice
  E-prime software will be used to determine the percentage accuracy and response time in seconds to a six separate cognitive challenges
Insulin sensitivity | After 2 weeks active juice and after 2 weeks placebo juice
  A hyperinsulinemic isoglycaemic clamp will be used to determine the amount of glucose required to maintain isoglycaemia (mg/kg/min)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Gilchrist, MB ChB, PhD, Principal Investigator — University of Exeter
Locations (1):
- NIHR Exeter Clinical Research Facility, Exeter, Devon, United Kingdom